CLINICAL TRIAL: NCT02697396
Title: A Randomized Controlled Trial of a Social Marketing Campaign to Increase HPV Vaccination Among Mexican American Children
Brief Title: Trial of a Social Marketing Campaign to Increase HPV Vaccination Among Mexican American Children
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The City College of New York (Other); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-069
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: HPV Vaccination
Keywords: Social Marketing Campaign; Mexican American Children; 16-069

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

GROUPS / COHORTS (2):
- with text messaging reminder system: Participants randomly assigned to the text messaging group will receive a text message reminding them of their child's vaccination eligibility once a week, starting one week after exposure to the social marketing campaign and time of consent.
  Interventions: Behavioral: Assessments; Other: Text Message Reminder
- without text messaging reminder system: Participants in this arm will receive no additional vaccination reminders. However, the study staff will ask and record if the participant's pediatrician provides appointment reminder cards, emails and/or calls prior to each scheduled vaccination as captured in the Outcomes Survey.
  Interventions: Behavioral: Assessments; Other: No Text Messaging

INTERVENTIONS:
Behavioral: Assessments — All participants, after consent, will be asked to complete the study contact form and then complete a baseline assessment with the RSA. This baseline assessment will take approximately 5 minutes.
Other: Text Message Reminder — Participants randomly assigned to the text messaging group will receive a text message reminding them of their child's vaccination eligibility once a week, starting one week after exposure to the social marketing campaign and time of consent.
  Groups: with text messaging reminder system
Other: No Text Messaging — Participants in this arm will receive no additional vaccination reminders.
  Groups: without text messaging reminder system

SUMMARY:
This project aims to raise awareness and improve HPV vaccination rates among children of Mexican American parents through the implementation of a tailored social marketing campaign which includes text messaging reminders.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will assess a social marketing campaign on HPV vaccination with and without a text messaging reminder system targeting Mexican Americans in a community-based setting, at the Ventanilla De Salud (Health Window, VDS) program and the Consulate on Wheels-Ventanilla De Salud Movil (Mobile Health Window, VDS on wheels) program of the Mexican Consulate. Investigators plan on recruiting 200 Mexican American parents of children ages 9 through 17. Every VDS attendee eligible for the study and who is willing to consent to participate will be invited to the study. Consenting participants will be randomized to either a follow-up reminder text messaging system or to the group which will not receive the text messaging reminders. All participants, regardless of text messaging arm, will evaluate the campaign and investigators will assess adherence to the HPV vaccine for the total sample.

ELIGIBILITY:
Inclusion Criteria:

* Born in Mexico or born in the U.S. but self-describes as Mexican-American Spanish is her/his primary language
* Has a minimum of one child between the ages of 9 and 17 who has not received the HPV vaccine and who lives with the parent/guardian as per self report
* Self-identifies as the child's main caregiver
* Currently owns a cell phone, uses text messaging services and is willing to accept text messages for this study

Exclusion Criteria:

* Will not be in the NYC area for the duration of the study period (6-9 months)
* Presence of a serious psychiatric or cognitive impairment likely to preclude meaningful informed consent and adherence to the protocol per the consenting professional's judgment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All recruitment will be completed by the MSKCC recruiting RSA who will approach all those attending the VDS at the Mexican Consulate in NYC and who are exposed to the social marketing campaign.
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete 3 doses of the HPV vaccine | 6 months
  This study will determine the effect of a social marketing campaign on HPV vaccination targeting Mexican American parents or guardians of vaccine-eligible children comparing the campaign alone against the campaign plus text message reminders on the proportion of participants who complete 3 doses of the HPV vaccine for their youngest eligible child.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Consulate General of Mexico in New York, New York, New York, United States

REFERENCES:
- [Derived] Aragones A, Gany F, Kaplan A, Bruno D. An opportunity to increase human papillomavirus vaccination rates: Change the guidelines. Hum Vaccin Immunother. 2022 Nov 30;18(6):2136444. doi: 10.1080/21645515.2022.2136444. Epub 2022 Oct 25. PMID 36282533
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT02697396/ICF_000.pdf